CLINICAL TRIAL: NCT00093834
Title: A Phase I Vaccine Safety and Chemotherapy Dose-Finding Trial of an Allogeneic GM-CSF-Secreting Breast Cancer Vaccine Given in a Specifically Timed Sequence With Immunomodulatory Doses of Cyclophosphamide and Doxorubicin
Brief Title: Vaccine Therapy With or Without Cyclophosphamide and Doxorubicin in Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0085 CDR0000391826; R01CA093714 (NIH); P30CA006973 (NIH); JHOC-J0085; JHOC-RPN-01012502; JHOC-RAC-0304-578
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin

INTERVENTIONS:
Biological: allogeneic GM-CSF-secreting breast cancer vaccine — The first three patients will receive a dose of 5 X 107 cells, and the next three will receive a dose of 5 X 108 cells. Then, if these two doses of vaccine alone are found to be safe, a fixed vaccine dose of 5 X 108 cells will be tested in combination with chemotherapy based on the safety of the allogeneic breast vaccine alone and the safety and bioactivity of a dose of 5 X 108 cells in the allogeneic pancreatic vaccine trial
Drug: cyclophosphamide — This trial will be a dose ranging study of a fixed sequence of drug doses in a three by three factorial matrix modeled after the theories of Plackett and Burman (Plackett et al., 1946), and is designed to determine the doses of CY and DOX that maximize the immunologic response to vaccination
Drug: doxorubicin hydrochloride — This trial will be a dose ranging study of a fixed sequence of drug doses in a three by three factorial matrix modeled after the theories of Plackett and Burman (Plackett et al., 1946), and is designed to determine the doses of CY and DOX that maximize the immunologic response to vaccination

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide and doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with cyclophosphamide and doxorubicin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cyclophosphamide and doxorubicin when given with vaccine therapy in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of vaccination comprising allogeneic sargramostim (GM-CSF)-secreting breast cancer cells with or without immunomodulation using cyclophosphamide and doxorubicin in women with stage IV breast cancer.
* Determine the doses of cyclophosphamide and doxorubicin that maximize vaccine-induced immunity, in terms of immune response to HER2/neu, in patients treated with these regimens.
* Compare in vivo immune response induced by these regimens, as measured by immunohistochemical analysis of vaccine site biopsies from these patients, with responses seen in prior preclinical and clinical studies.

Secondary

* Determine the time to disease progression in patients treated with these regimens.

OUTLINE: This is a dose-finding study.

The first 6 patients receive 1 of 2 doses of vaccine comprising allogeneic sargramostim (GM-CSF)-secreting breast cancer cells intradermally (ID) on day 0. Subsequent patients receive cyclophosphamide IV on day -1, vaccine at the higher dose ID on day 0, and doxorubicin IV on day 7. Treatment in all patients repeats every 4-6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after the third course receive a fourth course of treatment at approximately 4 months after completion of the third course.

Cohorts of 2-3 patients receive a fixed dose of vaccine in combination with escalating doses of doxorubicin and cyclophosphamide. Doses of cyclophosphamide and doxorubicin are escalated until an optimal dose of combination chemotherapy with a fixed dose of vaccine is achieved.

Patients are followed at 1 month and 4 months after completion of study therapy and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage IV disease
* Stable disease for ≥ 28 days
* Measurable or evaluable disease OR no evidence of disease
* Not eligible for potentially curative therapy
* Adequately treated CNS metastases are allowed
* Hormone receptor status:

  * Not specified
* HER-2/neu status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL (unless due to Gilbert's syndrome)
* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN

Renal

* Creatinine < 2.0 mg/dL

Cardiovascular

* Ejection fraction ≥ 45% by echocardiogram or MUGA

Pulmonary

* Asthma or chronic obstructive pulmonary disease allowed provided daily systemic corticosteroid therapy is not required

Immunologic

* No active autoimmune disease requiring systemic immunosuppressive therapy, including any of the following:

  * Inflammatory bowel disease
  * Systemic vasculitis
  * Scleroderma
  * Psoriasis
  * Multiple sclerosis
  * Hemolytic anemia
  * Immune-mediated thrombocytopenia
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Sjögren's syndrome
  * Sarcoidosis
  * Other rheumatologic disease
* HIV negative
* No active acute or chronic infection
* No allergy to corn

Other

* No other malignancy within the past 5 years except carcinoma in situ of the cervix, superficial nonmelanoma skin cancer, or superficial bladder cancer
* No active major medical or psychosocial problem that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy
* No other concurrent biologic therapy, including trastuzumab (Herceptin®)

Chemotherapy

* Prior adjuvant chemotherapy allowed
* Prior doxorubicin and cyclophosphamide allowed

  * Prior doxorubicin dose combined with planned study therapy dose must not exceed a lifetime cumulative dose of ≥ 450 mg/m^2
* More than 28 days since prior systemic chemotherapy
* No other concurrent systemic chemotherapy

Endocrine therapy

* More than 28 days since prior systemic corticosteroids
* Concurrent hormonal or endocrine therapy allowed

  * No concurrent systemic corticosteroids

Radiotherapy

* More than 28 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 28 days since prior participation in another investigational drug trial
* No other concurrent investigational drugs
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Toxicity of vaccine w/ & w/o cyclophosphamide+doxorubicin by history and phys. exam. at 28-42 days after each vaccination, 56-84 days after third vaccination, 6 months after first vaccination, and annually after first vaccination | 4 years
Toxicity of vaccine w/ & w/o cyclophosphamide+doxorubicin by CBC w/ differential at days 7, 14, 21, and 28-42 days after each vaccination, 56-84 days after third vaccination, 6 months after first vaccination, and annually after first vaccination | 4 years
Toxicity of vaccine w/ & w/o cyclophosphamide+doxorubicin by comprehensive metabolic panel at day 7 and 28-42 days after each vaccination, 56-84 days after third vaccination, 6 months after first vaccination, and annually after first vaccination | 4 years
Immune resp. of HER-2/neu by serum antibody titers, delayed hypersensitivity to HER-2/neu-derived peptides, and CD4+ T-cell resp. by ELISPOT at days 28-42 after each vaccination and days 56-84 after third vaccination | 4 years
Immune responses by immunohistochemical analysis of vaccine site biopsies at days 3 and 7 after the first and third vaccinations | 4 years

SECONDARY OUTCOMES:
Time to disease progression by history and physical examination, computed tomography, bone scans, and tumor markers as appropriate at days 28-42 after third and fourth vaccinations and days 56-84 after third vaccination | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Leisha A. Emens, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Emens LA, Armstrong D, Biedrzycki B, Davidson N, Davis-Sproul J, Fetting J, Jaffee E, Onners B, Piantadosi S, Reilly RT, Stearns V, Tartakovsky I, Visvanathan K, Wolff A. A phase I vaccine safety and chemotherapy dose-finding trial of an allogeneic GM-CSF-secreting breast cancer vaccine given in a specifically timed sequence with immunomodulatory doses of cyclophosphamide and doxorubicin. Hum Gene Ther. 2004 Mar;15(3):313-37. doi: 10.1089/104303404322886165. No abstract available. PMID 15018740